CLINICAL TRIAL: NCT04232644
Title: A Pilot, Randomized, Double-Blind, Active-Controlled, 2-Treatment, Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Abuse Liability of Dextroamphetamine Sulfate From an Abuse-Deterrent Immediate-Release Formulation (ADAIR)
Brief Title: Pilot Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Abuse Liability of an Abuse-Deterrent Immediate-Release Formulation (ADAIR)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vallon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAL-103
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: ADHD; Narcolepsy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Narcolepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Active Comparator): crushed d-amphetamine IR tablets
  Interventions: Drug: ADAIR 10mg IR capsules; Drug: Crushed d-amphetamine sulfate IR tablets
- Treatment B (Experimental): manipulated ADAIR IR capsules
  Interventions: Drug: ADAIR 10mg IR capsules; Drug: Crushed d-amphetamine sulfate IR tablets

INTERVENTIONS:
Drug: ADAIR 10mg IR capsules — manipulated ADAIR IR 3x10 mg capsules
Drug: Crushed d-amphetamine sulfate IR tablets — crushed d-amphetamine sulfate IR 6 x 5 mg tablets

SUMMARY:
This is a pilot randomized, double-blind, active-controlled, 2-treatment, crossover study to evaluate the PK, user experience and abuse liability of manipulated ADAIR compared to a manipulated commercially-available d-amphetamine sulfate IR formulation administered intranasally in non-dependent recreational stimulant users. The study is comprised of 4 phases: Screening, Qualification, Treatment, and Follow-up/Early Termination.

DETAILED DESCRIPTION:
VAL-103 is a phase 1, pilot, randomized, double-blind, active-controlled, 2-treatment crossover study. The study objectives include assessing the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of manipulated ADAIR 30 mg compared to crushed d-amphetamine sulfate IR 30 mg (DEX) administered IN in non-dependent recreational stimulant users. The primary PD endpoint is mean maximum drug liking (Emax) on a bipolar 100mm visual analog scale.

A total of 16 qualified subjects demonstrating a confirmed positive response to stimulants will enter the treatment phase. Safety will be assessed via adverse events, vital signs, ECGs, clinical laboratory tests, and Columbia Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
Inclusion Criteria:

* BMI within 18.5-32.0 kg/m2 and min weight of 50.0 kg
* healthy, according to med history, ECG, vital signs, lab results and physical exam
* clinical lab values within acceptable lab test range, unless otherwise deemed acceptable by PI
* SBP between 95-140 mmHg and DBP between 55-90 mmHg and HR between 50-100 bpm unless deemed not clinically significant by PI
* current or history of stimulant use for recreational purposes at least 10 times in lifetime and used stimulants at least once in the 12 weeks before screening
* experience with intranasal drug use for the purpose of recreational use on at least 3 occasions in the year prior to Screening
* ability to fast for at least 12 hours and consume standard meals
* agree not to have tattoo or body piercing until end of study
* female subject must be non-pregnant and non-lactating and fulfill at least one of following: participant is of childbearing potential and had used one of accepted contraception regimens from at least 30 days prior to first study drug and agrees to use two acceptable contraceptive regiment through at least 30 days after last dose of study drug or participant is of non-childbearing potential, defined as surgically sterile or is in a postmenopausal state
* a male subject must have met one of the following: participant is able to procreate and agreed to use one of accepted contraceptive regimens and not donate sperm from first study drug administration to at least 90 days after last drug administration or participant is unable to procreate, defined as surgically sterile and agreed to use a male condom from first study drug administration to at least 90 days after last drug administration

Exclusion Criteria:

* substance or alcohol dependence within the past 2 years
* history or presence of clinically significant abnormality as assessed by physical exam, med history, ECGs, vital signs, or lab results which in the opinion of the investigator would jeopardize the safety or the subject or validity of the study results
* history or presence of cardiovascular disorder, pre-existing structural cardiac abnormalities or other serious cardiac problems, prolonged QT syndrome, and associated risk factors
* abnormalities in the intranasal cavity or any condition that in the opinion of the PI would interfere with study procedures, data integrity, or compromise the safety of the subjects
* history or presence of mechanical gastrointestinal obstruction or any disease/conditions that affect bowel transit
* documented history of, or currently active, seizure disorder or history of clinically significant head injury or syncope of unknown origin
* history or presence of any psychiatric or neurological condition that, in the opinion of the PI, could get exacerbated by study drug exposure or interfere with study procedures
* subject with history of suicidal ideation or suicidal behavior as assessed by the Columbia Suicide Severity Rating Scale
* heavy smoker (>20 cigarettes per day) and/or is unable to abstain from smoking for a least 6 hours during the in-clinic periods
* history of severe allergic reaction to any substance, severe bronchial asthma, chronic obstructive airway, or previous status asthmaticus
* history of allergy or hypersensitivity to amphetamine salts, its excipients, or related substances
* history of food allergies, including lactose, and/or presence of any dietary restrictions
* positive test results for any of the following: HIV, Hep B, Hep C, positive drug screen at admission to the Qualification Phase or Treatment Phase, breath alcohol test and positive pregnancy test for females
* evidence of clinically significant hepatic or renal impairment including ALT or AST>1.5x the upper limit of normal (ULN) or bilirubin >1xULN
* known history or presence of: seizures or risk of seizure; tics or Tourette's Syndrome; psychosis, mania, bipolar disorder, suicidality or violent behavior; hyperthyroidism; Raynaud's Phenomenon; eye disorders
* individuals who have donated 50-499 mL of blood in the previous 30 days; or 500 mL or more in the previous 56 days
* donation of plasma by plasmapheresis within 7 days prior to first study drug administration
* difficulty with venous access or unsuitable or unwilling to undergo catheter insertion
* treatment with investigational drug within 5 times the elimination half-life, if known, or within 30 days prior to first drug administration or is concurrently enrolled in any research judged not to be scientifically or medically compatible with the study
* use of any prescription medication within 14 days prior to first study drug administration
* use of any OTC medications within 14 days prior to first study drug administration
* use of any prescription drugs, including MAO inhibitors, selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, triptans, tricyclic antidepressants, fentanyl, lithium, buspirone, St. Johns Wort and all medications which are cytochrome P450 (CYP450) 2D6 inhibitors in the 30 days or 5 half-lives (whichever was longer) prior to first study drug administration
* use of any alkalinizing agents within 30 days prior to first study drug administration
* individuals having undergone any major surgery within 6 months prior to start of study, unless deemed not clinically significant by PI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse event reporting | Day 1 to Day 9 (Treatment Phase)
  Assess the safety and tolerability as measured by the incidence, frequency, and severity of treatment-emergent adverse events
Abnormal Vital Signs | Day 1 to Day 9 (Treatment Phase)
  Number and percent of subjects with abnormal vital sign values
Abnormal ECG Values | Day 1 to Day 9 (Treatment Phase)
  Number and percent of abnormal ECG values
Abnormal clinical laboratory results | Day 1 to Day 9 (Treatment Phase)
  Number and percent of abnormal clinical laboratory results

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 24 hours post dose
  Maximum plasma concentration
Time to Maximum Plasma Concentration (tmax) | Up to 24 hours post dose
  Time to maximum plasma concentration
Area Under the Plasma Concentration AUC0-1h | Up to 24 hours post dose
  Area under the plasma concentration vs time curve from time 0 to 1 hour (AUC 0-1h)
Area Under the Plasma Concentration AUC0-2h | Up to 24 hours post dose
  Area under the plasma concentration vs time curve from time 0 to 2 hours (AUC0-2h)
Area Under the Plasma Concentration AUC0-4h | Up to 24 hours post dose
  Area under the plasma concentration vs time curve from time 0 to 4 hours (AUC0-4h)
Area Under the Plasma Concentration AUCt | Up to 24 hours post dose
  Area under the plasma concentration vs time curve from time 0 to the time of the last measurable concentration, or last sampling time t (AUCt)
Area Under the Plasma Concentration AUCinf | Up to 24 hours post dose
  Area under the plasma concentration vs time curve extrapolated to infinity (AUCinf)
Abuse quotient (AQ) | Up to 24 hours post dose
  Abuse quotient (AQ): Cmax/tmax
Terminal elimination rate constant λz | Up to 24 hours post dose
  Terminal elimination rate constant (λz)
Terminal elimination half-life t½ | Up to 24 hours post dose
  Terminal elimination half-life (t½)
Bipolar Ease of Snorting visual analog scale (VAS) | Up to 24 hours post dose
  Bipolar Ease of Snorting VAS minimum (peak) effect (Emin)
Bipolar Likeability of Snorting VAS | Up to 24 hours post dose
  Bipolar Likeability of Snorting VAS -minimum (peak) effect (Emin), maximum (peak) effect (Emax), time-averaged area under the effect curve from time 0 to 24 hours postdose (TA_AUE)
Bipolar Comfort of Snorting VAS | Up to 24 hours post dose
  Bipolar Comfort of Snorting VAS - minimum (peak) effect (Emin), maximum (peak) effect (Emax), time-averaged area under the effect curve from time 0 to 24 hours postdose (TA_AUE)
Subject-Rated Assessment of Intranasal Irritation (SRAII) | Up to 24 hours post dose
  Subject-Rated Assessment of Intranasal Irritation (SRAII) - maximum (peak) effect (Emax)and TEmax: time to maximum effect)
Percent of dose insufflated | 0 min (dosing time)
  Percent of dose insufflated

OTHER OUTCOMES:
Abuse Liability | Up to 24 hours post dose
  Abuse liability parameters measured by Visual Analogue Scales (VAS)
Subjective Drug Value Assessment | Up to 24 hours post dose
  Assessment of subjective drug value up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Whitaker, MD, Study Director — Vallon Pharmaceuticals, Inc.
Locations (1):
- BioPharma Services Inc., Toronto, Ontario, Canada